CLINICAL TRIAL: NCT06643936
Title: E3 Diabetes - Closing the Gap in Diabetes Control
Acronym: E3Diabetes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 24062508
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; self-monitoring; adherence; social determinants of health; health care system trust
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetes Team-Based Group (Experimental): A multidisciplinary team composed of a pharmacist, social worker, community health worker, and dietician will provide glucose monitoring, medication titration, diet education and reinforcement, and referrals for social needs. The pharmacist will remind patients to get A1C readings at 3 months and 6 months. The team will interact with the patients predominantly via tele-health remotely for 6 months.
  Interventions: Behavioral: E3 Multidisciplinary Team
- Diabetes Self-Guided Group (Active Comparator): A registered nurse will ensure patients have glucose monitors and supplies on enrollment and will call to remind patients to obtain A1C readings at 3 months and 6 months. Patients will continue with standard clinical care for type 2 diabetes in addition to receiving timed, mailed educational materials on type 2 diabetes monitoring and diabetes diet and lifestyle recommendations for 6 months.
  Interventions: Behavioral: E3 Self-Guided Type 2 Diabetes Education

INTERVENTIONS:
Behavioral: E3 Multidisciplinary Team — The E3 Multidisciplinary team is composed of a remote pharmacist, social worker, community health worker, and dietician working together to overcome barriers to diabetes control via behavioral change, medication adherence and titration, diet and lifestyle education and resource referrals for social needs.
  Arms: Diabetes Team-Based Group
Behavioral: E3 Self-Guided Type 2 Diabetes Education — Patients will receive timed, mailed educational materials on diabetes monitoring, diet and lifestyle modifications to supplement usual clinic based type 2 diabetes care with their primary care doctor. A registered nurse will ensure patients have glucometers and supplies, and remind patients to obtain A1C readings at 3 months and 6 months via phone call.
  Arms: Diabetes Self-Guided Group

SUMMARY:
This study aims to decrease the racial gap in type 2 diabetes control in African American and Latinx patients in Rush University Medical Center clinics.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of death in the US as well as in Chicago. Risk factors for CVD include hypertension, diabetes, and lifestyle factors such as smoking, diet, and obesity. Among the critical social and structural determinants of cardiovascular health are food access, neighborhood safety, education, poverty, and chronic stress. Chicago and its surrounding region suffer from longstanding racial disparities in both social conditions and chronic disease burden, contributing to stark racial gaps in cardiometabolic disease mortality. Life expectancy is as high as 84 years on Chicago's North Side, but only 68 years on the West Side - a gap of 16 years. Cardiometabolic disease accounts for 40 to 50% of this lifespan gap. The diabetes-related death rate is 70% higher among Chicago's African Americans than among non-African Americans. In Rush primary care clinics, under conditions of usual clinical care, African American and Latinx patients with diabetes have worse glycemic control than white patients, raising the question whether modifying the model of diabetes care from intermittent clinic-based care to more frequent home-based care remote monitoring might reduce these stubborn disparities. We are proposing a feasibility trial of a remote diabetes monitoring, social care, medication adherence and dietary intervention to improve diabetes control among African American and Latinx patients attending primary care clinics at Rush University Medical Group locations with the eventual aim of closing the racial/ethnic disparity in diabetes control. The proposed feasibility trial will use a randomized-control, four-pronged approach to improve glycemic control. The intervention group will receive the following: 1) remote glucose monitoring, 2) a multidisciplinary team to address social needs, 3) medication titration and adherence support, and 4) culturally tailored diabetes self-management and dietary education. The control group will receive standard of care diabetes primary care in addition to dietary education around diabetes through written materials. We hypothesize that E3 Diabetes program participants will achieve a change in A1c of 0.5 in at least 30% of the participants in 6 months, and will be a greater percentage than seen with the propensity matched control of African American and Latinx patients receiving usual care for Diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years and older
* African American and/or Latinx
* Uncontrolled Type 2 Diabetes, A1C >/= 8.0 within the last 3 months
* Following with Rush primary care provider in eligible Rush primary care clinics
* Access to cellphone

Exclusion Criteria:

* Patient has Type 1 Diabetes
* Patient is already participating in another remote diabetes monitoring program
* Patient is not interested in participating in the program
* Patient has already participated in the E3 hypertension program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1C | baseline, 6 months, 12 months
  We hypothesize that the E3 Multidisciplinary team group patients will achieve a change in A1c of 0.5 in at least 30% of participants in 6 months compared to baseline, and this will be a greater percentage than seen with Self-guided group of African American and Latinx patients receiving usual care for Diabetes with educational materials. A1C will be measured at 12 months to check for persistence in A1C improvement as compared to 6 months and baseline.

SECONDARY OUTCOMES:
Health Care System Distrust | 6 months and 12 months
  To test the hypothesized mechanisms of change of the intervention by assessing the relationship between change in the following intervening behavioral targets and change in glycemic control at 6 and 12 months: perceived trust in healthcare system
Diabetes Self Management | 6 months and 12 months
  To test the hypothesized mechanisms of change of the intervention by assessing the relationship between change in the following intervening behavioral targets and change in glycemic control at 6 and 12 months: diabetes self management skills (e.g. monitoring blood glucose levels, food intake, physical activity)
Medication Adherence | 6 months and 12 months
  To test the hypothesized mechanisms of change of the intervention by assessing the relationship between change in the following intervening behavioral targets and change in glycemic control at 6 and 12 months: daily medication adherence
Primary Care Visit Attendance | 6 months and 12 months
  To test the hypothesized mechanisms of change of the intervention by assessing the relationship between change in the following intervening behavioral targets and change in glycemic control at 6 and 12 months: attending primary care visits at 3 and 6 months after enrollment.

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Individual patient data will not be shared, however aggregate patient data may be shared with other researchers

DOCUMENTS (1):
  • Informed Consent Form (2024-10-10): https://cdn.clinicaltrials.gov/large-docs/36/NCT06643936/ICF_000.pdf